CLINICAL TRIAL: NCT03289442
Title: Impact of Supine Position on Colonoscopy Insertion: a Randomized Controlled Trial
Brief Title: Supine Position for Colonoscopy Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: No.85 Hospital, Changning, Shanghai, China (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director, Head of Department of Gastroenterology, Principal Investigator, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: position-2
Record Dates: First submitted 2017-09-17; First posted 2017-09-21 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Colonoscopy Insertion; Patient Position
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supine position group (Experimental)
  Interventions: Procedure: supine position
- left lateral position (No Intervention)

INTERVENTIONS:
Procedure: supine position — patients were positioned on their supine position to receive colonoscopy insertion
  Arms: supine position group

SUMMARY:
The purpose of this study is to determine whether the supine position is better than the left lateral horizontal body position to decrease cecal intubation time, patients' pain and the difficulty of colonoscopy insertion.

DETAILED DESCRIPTION:
Left lateral position is conventionally performed to initiate colonoscopy, yet no evidence has demonstrated its efficacy and advantages. Left lateral position for insertion, which results in air rising away from the left colon and producing acute bends in the sigmoid,might increase the risk of colonoscopy loop formation.When there is difficulty advancing the colonoscope, supine position can be employed to ensure cecal intubation. Therefore, we perform a randomized controlled trial to compares supine position with left lateral position for the safety and efficacy of colonoscopy insertion.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18-75 years
2. underwent screening, surveillance, and diagnostic colonoscopy

Exclusion Criteria:

1. <18 or >75 years old
2. major psychiatric disorders, colonic resection, pregnancy, presence of any contraindications for colonoscopy (eg, severe heart failure, renal insufficiency)
3. Patients with severe cardiopulmonary and renal disease
4. Patients who are unwilling or unable to consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
cecal intubation time | 2 hour
  Cecal intubation time is the insertion time taken from first visualization of rectal mucosa to cecum and cecal intubation was confirmed by identifying the characteristic anatomical landmarks of the triradiate fold, appendiceal orifice, and ileocecal valve.

SECONDARY OUTCOMES:
descending colon intubation time | 1 hour
  Descending colon intubation time is the insertion time taken from first visualization of rectal mucosa to descending colon and descending colon was identified by the presence of straight colonic lumen and affirmed by an independent observer simultaneously.
patients' pain score | 3 hour
  patients' discomfort will be assessed by a 10-cm visual analog scale, in which a score of 0 denoted no pain and a score of 10 denoted unbearable pain
patients' acceptance to unsedated or sedated colonoscopy in the future screening or examination | 3 hour
  when colonoscopy insertion is completed, patients will be asked whether they would accept similar unsedated or sedated colonoscopy in the future screening or examination

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Willcock H, Gold DM. Supine Colonoscopy: An Advantage over Left Lateral in Synchronous Proctological Surgery. J Laparoendosc Adv Surg Tech A. 2016 Jun;26(6):475-7. doi: 10.1089/lap.2015.0609. Epub 2016 Mar 16. PMID 26982385
- [Result] Waye JD, Yessayan SA, Lewis BS, Fabry TL. The technique of abdominal pressure in total colonoscopy. Gastrointest Endosc. 1991 Mar-Apr;37(2):147-51. doi: 10.1016/s0016-5107(91)70673-1. PMID 2032597
- [Derived] Zhao S, Yang X, Meng Q, Wang S, Fang J, Qian W, Xia T, Pan P, Wang Z, Gu L, Chang X, Zou D, Li Z, Bai Y. Impact of the supine position versus left horizontal position on colonoscopy insertion: a 2-center, randomized controlled trial. Gastrointest Endosc. 2019 Jun;89(6):1193-1201.e1. doi: 10.1016/j.gie.2019.01.009. Epub 2019 Jan 18. PMID 30660634